CLINICAL TRIAL: NCT06381167
Title: Endoscopic Bi-portal Decompression Versus Microscopic Decompression in Cases of Lumbar Canal Stenosis
Brief Title: Endoscopic Decompression Versus Microscopic Decompression in Lumbar Canal Stenosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Soliman Ali Noman, doctor, Assiut University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Endoscopic decompression
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Endoscopic bi-portal decompression; Microscopic decompression; Lumbar canal stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic bi-portal decomprssion (Experimental): patients with lumbar canal stenosis will undergo endoscopic decompression
  Interventions: Procedure: Endoscopic Decompressive Laminectomy
- Microscopic decompression (Experimental): patients with lumbar canal stenosis will undergo microscopic decompression
  Interventions: Procedure: Endoscopic Decompressive Laminectomy

INTERVENTIONS:
Procedure: Endoscopic Decompressive Laminectomy — the patients will undergo block randomization for either endoscopic or microscopic decompression
  Other Names: Microscopic Decompressive Laminectomy

SUMMARY:
To compare between the clinical and surgical efficacies of bi-portal endoscopic and microscopic decompressive laminectomy in patients with degenerative lumbar spinal stenosis.

DETAILED DESCRIPTION:
Lumbar canal stenosis is a disease caused by the compression of the dural sac and nerve root due to various factors such as hypertrophy of the ligamentum flavum (LF), facet joint hypertrophy, disc herniation, and spondylolisthesis, resulting in low back pain, leg pain with or without numbness, intermittent claudication, and bladder and bowel dysfunction in which intermittent neurogenic claudication is the main feature (1, 2).

Traditional surgical approaches include open laminotomy decompression, foraminotomy, discectomy, and fusion. Conventional open lumbar decompression has a long history and has the advantages of adequate decompression and clear visualization of neural structures, while surgical invasiveness and extensive stripping of paraspinal muscles and soft tissues may lead to a series of problems such as postoperative low back pain, spinal instability, and prolonged hospital stay and time to return to normal life after the operation (3).

Minimally invasive spine surgery has become increasingly popular in recent years. Unilateral bi-portal endoscopy (UBE) was proposed by Heo in 2017 to treat degenerative lumbar spinal diseases with less damage to the paraspinal muscles (4).

Minimally invasive decompression was introduced as a tissue-sparing alternative and applied to lumbar central stenosis. Minimally invasive decompression revealed good clinical outcomes comparable to those of conventional surgery (5, 6). It also showed a reasonable operative time, shorter hospital stay, and reduced blood loss, time to mobilization, postoperative pain, and narcotic use when compared to that seen with conventional surgery (7).

However, it presents some disadvantages, including poor visualization, difficulty of instrument manipulation, potential to induce inadequate decompression, and longer operative time than other minimally invasive surgeries (8).

ELIGIBILITY:
Inclusion Criteria:

* Patients with acquired degenerative lumbar canal stenosis. Age >40 years. Single or Double level stenosis

Exclusion Criteria:

* Post-traumatic lumbar canal stenosis. Previous spine surgery. Multi-level stenosis more than 2 levels. Associated instability e.g. spondylolisthesis. Spinal diseases (e.g., ankylosing spondylitis, infection, spine tumor, fracture, or neurologic disorders).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index ODI scores for low back pain and neuropathic pain | one year
  3,6 and 12-month follow-up after surgery

SECONDARY OUTCOMES:
visual analog scale (VAS) score for low back and lower extremity radiating pain | one year
  3,6 and 12-month follow-up after surgery
European Quality of Life-5 Dimensions (EQ-5D) score | one year
  3,6 and 12-month follow-up after surgery
painDETECT score | one year
  3,6 and 12-month follow-up after surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park SM, Park J, Jang HS, Heo YW, Han H, Kim HJ, Chang BS, Lee CK, Yeom JS. Biportal endoscopic versus microscopic lumbar decompressive laminectomy in patients with spinal stenosis: a randomized controlled trial. Spine J. 2020 Feb;20(2):156-165. doi: 10.1016/j.spinee.2019.09.015. Epub 2019 Sep 19. PMID 31542473
- [Background] Heo DH, Son SK, Eum JH, Park CK. Fully endoscopic lumbar interbody fusion using a percutaneous unilateral biportal endoscopic technique: technical note and preliminary clinical results. Neurosurg Focus. 2017 Aug;43(2):E8. doi: 10.3171/2017.5.FOCUS17146. PMID 28760038
- [Background] Wang X, Tian Z, Mansuerjiang M, Younusi A, Xu L, Xiang H, Cao L, Wang C. A single-arm retrospective study of the clinical efficacy of unilateral biportal endoscopic transforaminal lumbar interbody fusion for lumbar spinal stenosis. Front Surg. 2023 Jan 23;9:1062451. doi: 10.3389/fsurg.2022.1062451. eCollection 2022. PMID 36756660